CLINICAL TRIAL: NCT00643357
Title: Study of the Efficacy and Safety of KALINOX® 170 Bar for the Performance of Care Procedures in Children With Burns
Acronym: Burns
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patient recruited due to current guidelines for the pain related to burn
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-002698-38
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Burns
Keywords: children with burns; Child between 5 and 15 years of age , burned for many days and who has to undergo at least 3 procedures of care
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 50% Oxygen/50% Nitrous oxide premix (Kalinox® 170 bar)
  Interventions: Drug: 50% Oxygen/50% Nitrous oxide premix (KALINOX 170 bar)
- B (Placebo Comparator): 50%Oxygen/50% Nitrogen premix
  Interventions: Drug: 50%Oxygen/50% Nitrogen premix

INTERVENTIONS:
Drug: 50% Oxygen/50% Nitrous oxide premix (KALINOX 170 bar) — gaz flow between 4 to 15 L/min inhalation between 15 to 60 minutes
  Arms: A
Drug: 50%Oxygen/50% Nitrogen premix — inhalation between 15 to 60 minutes gaz flow between 4 to 15 l/min
  Arms: B

SUMMARY:
The purpose of this study is to assess the efficacy and the safety of Kalinox® 170 bar, over a period of three consecutive care procedures in burned children. It's a international (Spain, France, Tunisia and Belgium) study with 8 investigator centers.

DETAILED DESCRIPTION:
Pain due to burns is one of the most intense and persistent types of pain. This pain consists of a permanent background pain, overlaid by episodes of temporary exacerbations triggered by treatment procedures or burn-care procedures.

Care procedures, such as changing the dressings or cleaning the wounds, make it necessary to handle the painful areas, and this causes transient intense pain.

Analgesia with a 50/50 mix of nitrous oxide and oxygen is a simple and effective technique, which induces a state of light sedation during which verbal contact is not lost, which is rapidly reversible and is devoid of any major side effects. This gas is used in paediatrics for carrying out painful procedures of a short duration, such as lumbar puncture and minor surgery.

The nitrous oxide/oxygen mix has also been used to treat the pain induced by care procedures in children with burns for more than 30 years.

The objective of our study is to obtain qualitative and quantitative data about the efficacy of Kalinox® 170 bar in care procedures in children with burns.

ELIGIBILITY:
Inclusion Criteria:

* Child between 5 and 15 years of age , burned for many days and who has to undergo at least 3 procedures of care

  * potentially mildly to moderately painful
  * lasting for at least 15 minutes and for less than 30 minutes
  * eligible to receive short-term prophylactic analgesic treatment
  * for whom the consent form has been signed (parent and child)

Exclusion criteria:

* Child treated under general anaesthesia
* Child physically or mentally incapable of responding to an assessment of his/her pain on a visual scale.
* Child suffering from moderate to severe pain when beginning the care procedure (FPSr > 4)
* Exclusion criteria linked to the product

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The intensity of the pain was assessed using the "Faces Pain Scale Revised" | Faces Pain Scale Revised